CLINICAL TRIAL: NCT03712046
Title: Comparaison Entre la Performance du 18F-FDG PET/CT et de la Scintigraphie Osseuse/Gallium ou de la Scintigraphie Osseuse/Globules Blancs marqués /Souffre colloïdal Dans le Diagnostic d'Une ostéomyélite du Pied ou de la Cheville
Brief Title: Comparison of FDG PET and Bone Scintigraphy/Labelled Leukocyte/Gallium Scintigraphy in Diabetic Foot Osteomyelitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient recruitment
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18.200
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Foot Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): PET-CT imaging of the ankles and feet following injection of 18F-FDG
  Interventions: Diagnostic Test: 18F-FDG PET-CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET-CT — Patient will receive one injection of 18F-FDG and then undergo PET-CT imaging

SUMMARY:
Diabetic foot osteomyelitis is a common and serious complication of diabetes. While the diagnosis of soft tissue infection can be made with simple physical examination in most cases, bone involvement can be harder to diagnose, often requiring medical imaging. In addition to conventional radiological examinations (x-ray and MRI) nuclear medicine procedures can also provide important physiological information in these patients. These procedures include triple phase bone scan combined with Gallium scintigraphy or a combination of labelled leukocyte scintigraphy and bone marrow scintigraphy using sulfur colloid. These procedure, while they provide useful physiological information, are time consuming, generally requiring at least 2 separate image acquisition on separate days, and can be costly.

18F-FDG is a glucose analog that can be used for PET imaging. In addition to its application in oncology, the literature has shown that FDG can be used to investigate a wide variety of inflammatory and infectious conditions, including diabetic foot infections.

The aim of this study is to compare the usefulness of FDG PET imaging versus "conventional" nuclear medicine (either bone scan and Gallium scintigraphy or labelled leukocytes and sulfur colloid scintigraphy) in patient with suspected diabetic foot osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient with suspected diabetic foot osteomyelitis referred for nuclear medicine examination (bone scan and Gallium or labelled leukocytes).
* Being treated or followed by a physician at CHUM

Exclusion Criteria:

* Pregnant woman
* Breastfeeding patient
* Claustrophobia/patient unable to complete imaging procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of 18F-FDG PET-CT for the diagnosis of diabetic foot osteomyelitis | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada